CLINICAL TRIAL: NCT05750056
Title: Effect of Intraoperative Intravenous Lidocaine on the Quality of Recovery Following Colorectal Endoscopic Submucosal Dissection
Brief Title: Dose Systemic Lidocaine Improve the Quality of Recovery After Colorectal Endoscopic Submucosal Dissection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Clinical Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K2020-05-029-02
Record Dates: First submitted 2023-01-28; First posted 2023-03-01 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Recovery
Keywords: endoscopic submucosal dissection; lidocaine; cognitive recovery; quality of recovery
MeSH Terms: interventions — Lidocaine; Saline Solution; Sodium Chloride; Propofol; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Patients received an intravenous bolus injection of lidocaine 1.5 mg/kg over 10 min before induction of anesthesia, followed by a continuous infusion of 2 mg/kg/h until the end of the surgery.
  Interventions: Drug: lidocaine; Drug: Propofol; Drug: Sufentanil
- Placebo group (Placebo Comparator): Patients received a perioperative 0.9% saline infusion at the same rate as the lidocaine infusion.
  Interventions: Drug: 0.9% saline; Drug: Propofol; Drug: Sufentanil

INTERVENTIONS:
Drug: lidocaine — Patients received an intravenous bolus injection of lidocaine 1.5 mg/kg over 10 min before induction of anesthesia, followed by a continuous infusion of 2 mg/kg/h until the end of the procedure.
  Other Names: Lidocaine IV
  Arms: Lidocaine group
Drug: 0.9% saline — Patients received a perioperative saline infusion at the same rate and volume as the lidocaine infusion.
  Other Names: 0.9% sodium chloride
  Arms: Placebo group
Drug: Propofol — An i.v. bolus injection of propofol 1 mg/kg was given to all patients. Propofol was then titrated if necessary to produce unconsciousness during the introduction of the endoscope. Afterward, the anesthesiologist determined the dose of propofol and titrated to effect.
  Other Names: Propofol injection
Drug: Sufentanil — Sufentail 0.1 ug/kg was administered for sedation induction.
  Other Names: Sufentanil injection

SUMMARY:
Endoscopic submucosal dissection (ESD) is a common procedure that requires a long procedural time. Procedure Sedation is commonly provided to alleviate patients' discomfort and facilitate the implementation of procedures. We conducted a prospective study to determine the effect of intravenous infusion of lidocaine in the cognitive domain of the postoperative quality of recovery scale on day 3 after ESD.

DETAILED DESCRIPTION:
Colorectal cancer occurred in more than 1.9 million new cases and 935,000 deaths in 2020 and ranked third in incidence and second in mortality globally. Endoscopic submucosal dissection (ESD) is the current standard for treating large colorectal polyps and has been shown to reduce colorectal cancer-related mortality. Sedation is commonly provided to alleviate patients' discomfort and facilitate the implementation of procedures.

Lidocaine is an amide local anesthetic with analgesic, anti-hyperalgesic, and anti-inflammatory properties. Its safety in appropriate amounts has been established. The current evidence gap is whether the use of systematic lidocaine affects the quality of recovery after ESD. Thus, the aim of this study is to determine the effect of intravenous infusion of lidocaine in the cognitive domain of the postoperative quality of recovery scale on day 3 after ESD.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) classification I-III;
2. Scheduled for endoscopic colorectal mucosal dissection.

Exclusion Criteria:

1. Patient refuses to participate;
2. BMI greater than 30;
3. Allergic or contraindication to study drugs;
4. History of chronic pain and long-term use of analgesic medication;
5. Severe arrhythmia;
6. Hepatic and renal dysfunction;
7. Any other conditions precluded study inclusion, such as cognitive impairment, pregnancy, or inability to communicate in Mandarin Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive recovery | Day 3 postoperatively
  Postoperative cognitive recovery will be measured using the Postoperative Quality of Recovery Scale (PostopQRS). The PostopQRS is a multidimensional survey-based tool, which includes a domain designed to measure recovery in the cognitive domain of the PostopQRS over time during the postoperative period. The instrument is administered preoperatively to provide individual baseline measurements for each patient. Tests produce performance scores. Higher scores mean a better outcome. The recovery outcome is defined as returning to at least baseline values.

SECONDARY OUTCOMES:
Incidence of postoperative cognitive recovery | 30 minutes after endoscope removal
  Postoperative cognitive recovery will be measured using the Postoperative Quality of Recovery Scale (PostopQRS). The PostopQRS is a multidimensional survey-based tool, which includes a domain designed to measure recovery in the cognitive domain of the PostopQRS over time during the postoperative period. The instrument is administered preoperatively to provide individual baseline measurements for each patient. Tests produce performance scores. Higher scores mean a better outcome. The recovery outcome is defined as returning to at least baseline values.
Incidence of postoperative cognitive recovery | Day 1 postoperatively
  Postoperative cognitive recovery will be measured using the Postoperative Quality of Recovery Scale (PostopQRS). The PostopQRS is a multidimensional survey-based tool, which includes a domain designed to measure recovery in the cognitive domain of the PostopQRS over time during the postoperative period. The instrument is administered preoperatively to provide individual baseline measurements for each patient. Tests produce performance scores. Higher scores mean a better outcome. The recovery outcome is defined as returning to at least baseline values.
Incidence of postoperative cognitive recovery | Day 7 postoperatively
  Postoperative cognitive recovery will be measured using the Postoperative Quality of Recovery Scale (PostopQRS). The PostopQRS is a multidimensional survey-based tool, which includes a domain designed to measure recovery in the cognitive domain of the PostopQRS over time during the postoperative period. The instrument is administered preoperatively to provide individual baseline measurements for each patient. Tests produce performance scores. Higher scores mean a better outcome. The recovery outcome is defined as returning to at least baseline values.
Incidence of overall recovery | 30 minutes after endoscope removal
  The Postoperative Quality of Recovery Scale (PostopQRS) is a multidimensional survey-based tool, which contains physiological, emotive, nociceptive, activities of daily living, and cognitive recovery over time. Nociceptive, emotive, and activities of daily living that can be scored in a categorical fashion. In the cognitive domain, tasks receive a performance score. In the physiologic domain, values are transformed and categorized as acceptable, somewhat or far outside of the desirable boundaries, based on normative population data. Higher scores mean a better outcome, except for nociceptive domain. Overall recovery is postoperative values equaling or exceeding individual baseline values in each of the domains of the PostopQRS. The incidence of recovery is expressed as a percentage of participants recovered/group total at each time point.
Incidence of overall recovery | Day 1 postoperatively
  The Postoperative Quality of Recovery Scale (PostopQRS) is a multidimensional survey-based tool, which contains physiological, emotive, nociceptive, activities of daily living, and cognitive recovery over time. Nociceptive, emotive, and activities of daily living that can be scored in a categorical fashion. In the cognitive domain, tasks receive a performance score. In the physiologic domain, values are transformed and categorized as acceptable, somewhat or far outside of the desirable boundaries, based on normative population data. Higher scores mean a better outcome, except for nociceptive domain. Overall recovery is postoperative values equaling or exceeding individual baseline values in each of the domains of the PostopQRS. The incidence of recovery is expressed as a percentage of participants recovered/group total at each time point.
Incidence of overall recovery | Day 3 postoperatively
  The Postoperative Quality of Recovery Scale (PostopQRS) is a multidimensional survey-based tool, which contains physiological, emotive, nociceptive, activities of daily living, and cognitive recovery over time. Nociceptive, emotive, and activities of daily living that can be scored in a categorical fashion. In the cognitive domain, tasks receive a performance score. In the physiologic domain, values are transformed and categorized as acceptable, somewhat or far outside of the desirable boundaries, based on normative population data. Higher scores mean a better outcome, except for nociceptive domain. Overall recovery is postoperative values equaling or exceeding individual baseline values in each of the domains of the PostopQRS. The incidence of recovery is expressed as a percentage of participants recovered/group total at each time point.
Incidence of overall recovery | Day 7 postoperatively
  The Postoperative Quality of Recovery Scale (PostopQRS) is a multidimensional survey-based tool, which contains physiological, emotive, nociceptive, activities of daily living, and cognitive recovery over time. Nociceptive, emotive, and activities of daily living that can be scored in a categorical fashion. In the cognitive domain, tasks receive a performance score. In the physiologic domain, values are transformed and categorized as acceptable, somewhat or far outside of the desirable boundaries, based on normative population data. Higher scores mean a better outcome, except for nociceptive domain. Overall recovery is postoperative values equaling or exceeding individual baseline values in each of the domains of the PostopQRS. The incidence of recovery is expressed as a percentage of participants recovered/group total at each time point.
Propofol consumption | During the colonoscopy procedure
  Propofol consumption will be recorded during the colonoscopy procedure.
Endoscopitst satisfacrion | At completion of colonoscopy procedure
  Endoscopitst satisfacrion will be evaluated using a five-point Likert scale (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, and 1=very dissatisfied).
Patient satisfaction | On 1 day postoperatively
  Patient satisfaction will be evaluated using a five-point Likert scale (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, and 1=very dissatisfied).
Incidence of adverse events | Up to 24 hours postoperatively
  Adverse events such as bradycardia, tachycardia, hypertension, hypotension, and hypoxia will be recorded during the trial.

OTHER OUTCOMES:
Emergency time | Immediately after the colonoscopy completely withdrawn
  Emergency time is defined as the interval from the end of colonoscopy to the MOAA/S score equal to five.
Patient willingness to recommend screening | Day 1 postoperatively
  Patients will be asked whether they would recommend bronchoscopy screening to a friend or a relative (Yes/No/Unsure).
Patient willingness to repeat the procedure | Day 1 postoperatively
  Patients will be asked whether they would repeat the identical procedural process (Yes/No/Unsure)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zheng, MD, Study Chair — Fujian Provincial Hospital
Locations (1):
- Fujian provincial hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the individual deidentified participant data underlying published results, the study protocol, and the statistical analysis plan can be accessed upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We would like to share our IPD beginning 3 months following the publication of the main results.
Access Criteria: All of the individual participant data collected during the trial, the study protocol, the statistical analysis plan, and the clinical study report can be accessed with approval from the corresponding author.

REFERENCES:
- [Derived] Liang Y, Qian B, Zhuo Y, Zhang J, Gao W, Li H, Zhang X, Lin W. Intravenous Lidocaine and Cognitive Recovery After Endoscopic Submucosal Dissection: A Randomized Controlled Trial. Drug Des Devel Ther. 2025 Nov 22;19:10343-10355. doi: 10.2147/DDDT.S557688. eCollection 2025. PMID 41312048